CLINICAL TRIAL: NCT04336943
Title: Durvalumab (MEDI4736) and Olaparib (AZD2281) for Treatment of Biochemically Recurrent Prostate Cancer in Men Predicted to Have a High Neoantigen Load: A Multicenter Pilot Study
Brief Title: Durvalumab and Olaparib for the Treatment of Prostate Cancer in Men Predicted to Have a High Neoantigen Load
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Washington (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Michael Schweizer, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1007001; NCI-2020-01860 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10509 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Prostate Adenocarcinoma
MeSH Terms: interventions — durvalumab; Immunoglobulin G; Disulfides; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (durvalumab, olaparib) (Experimental): All patients receive durvalumab IV over 1 hour on day 1 of each cycle. Patients with CDK12 mutation and MMRd/MSI-high also receive olaparib PO BID on days 1- 28 of cycles 3-6. Patients with homologous recombination mutation also receive olaparib PO BID on days 1-28 of cycles 1-6. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Drug: Olaparib; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736; 1428935-60-7
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well durvalumab and olaparib work in treating prostate cancer in men predicted to have specific genetic mutations (a high neoantigen load). Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. PARPs are proteins that help repair DNA mutations. PARP inhibitors, such as olaparib, can keep PARP from working, so tumor cells can't repair themselves, and they may stop growing. Giving durvalumab and olaparib may kill more tumor cells in patients with prostate cancer predicted to have a high neoantigen load.

DETAILED DESCRIPTION:
OUTLINE:

All patients receive durvalumab IV over 1 hour on day 1 of each cycle, total 6 cycles. Starting cycle 4, patients with CDK12 mutations and mismatch repair deficiency (MMRd)/microsatellite instability (MSI)-high will also receive olaparib orally (PO) twice daily (BID) on days 1- 28 of cycles 4-6. Patients with homologous recombination mutation will also receive olaparib PO BID on days 1-28 of cycles 1-6. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 weeks, and then every 12 weeks to complete 24 months (at 9, 12, 15, 18, 21 and 24 months).

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of adenocarcinoma of the prostate
* The patient must have received definitive local therapy for prostate cancer, consisting of either radiation therapy and/or prostatectomy (salvage or adjuvant radiation post-prostatectomy is not exclusionary)
* PSA must be >= 2 ng/ml if received only prior definitive radiation (no PSA threshold required if prior prostatectomy was performed) with a PSA doubling time (PSADT) =< 10 months:

  * PSADT calculation must include all recorded PSA values > 0.2 ng/ml over the past 6 months prior to randomization, with a minimum of 3 values spaced at least 2 weeks apart, with each included value preferably measured at the same laboratory. PSA values obtained prior to localized therapy will be excluded
  * The calculation of PSADT is based on the natural log of PSA
* Prior salvage radiation or not a candidate for localized salvage radiation due to subject preference or clinical assessment based upon disease characteristics and/or subject co-morbidities
* Prior hormonal therapy (i.e. androgen deprivation therapy) when given as neoadjuvant/concurrent/adjuvant therapy along with definitive radiation is allowed, provided this was stopped >= 6 months prior to starting treatment per protocol AND testosterone is >= 150 ng/dl
* No evidence of metastatic disease on imaging by whole body bone scan and computed tomography (CT) or magnetic resonance imaging (MRI) of the chest/abdomen/pelvis within 6 weeks before study therapy start day. PSMA positron emission tomography (PET) or fluciclovine scan within 6 weeks of start day may substitute other imaging studies.

  * Patients with oligometastatic disease (i.e. =< 3 sites) detectable on advanced imaging only (e.g. PSMA or fluciclovine PET) are eligible
  * Abdominal or pelvic lymph nodes measuring =< 2 cm in short axis are allowed
* Biomarker positive:

  * Biallelic CDK12 inactivating mutations as documented using a clinical grade sequencing assay performed in a Clinical Laboratory Improvement Act (CLIA)/College of American Pathologists (CAP) certified laboratory or
  * MMRd/MSI-high as documented using a clinical grade assay performed in a CLIA/CAP certified laboratory or
  * Loss of function mutations in homologous recombination genes (i.e. homologous recombination deficiency; HRD) as documented using a clinical grade sequencing assay performed in a CLIA/CAP certified laboratory. Homologous recombination genes include, but not limited to BRCA1, BRCA2, ATM, CHEK2, PALB2, RAD51D, NBN, GEN1, RAD51C, MRE11A, BRIP11A, FAM175A.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Age > 18 years at time of study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Hemoglobin >= 10.0 g/dL with no blood transfusion in the past 28 days (within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) be >= 1.5 x 10^9/L (within 28 days prior to administration of study treatment)
* Platelet count >= 100 x 10^9/L (within 28 days prior to administration of study treatment)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to administration of study treatment). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be =< 5 x ULN (within 28 days prior to administration of study treatment)
* Patient must have creatinine clearance (CL) >= 51 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance (within 28 days prior to administration of study treatment)
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Patients must have a life expectancy >= 16 weeks
* Body weight > 30 kg
* Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential

Exclusion Criteria:

* Prior chemotherapy for prostate cancer, unless done in the neoadjuvant setting, and if the last dose was > 6 months prior to enrollment
* Any prior treatment with a PD1 or PD-L1 inhibitor, including durvalumab
* Any prior treatment with a PARP inhibitor, including olaparib
* History of another primary malignancy except for

  * Malignancy treated with curative intent and with no known active disease >= 3 years before the first dose of durvalumab and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis
* Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the treating physician (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, corrected QT interval by Fridericia [QTcF] prolongation > 470 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or olaparib may be included only after consultation with the study physician
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, extensive bilateral lung disease on high resolution computed tomography (HRCT) scan, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea or any psychiatric disorder that prohibits obtaining informed consent
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Immunocompromised patients, e.g., patients with uncontrolled human immunodeficiency virus (HIV). HIV+ patients will be allowed on the study if on highly active antiretroviral therapy (HAART) and disease is controlled: CD4 >= 350 cell/mcl, undetectable viral load, and no prophylactic (PPX) antibiotics

  * Note: HIV screening is not required to be eligible for this study
* Active infection including tuberculosis (TB testing only performed if deemed necessary per standard clinical practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the sponsor investigator
  * Patients with celiac disease controlled by diet alone
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab. Note: Patients, if enrolled, should not receive live vaccine whilst receiving durvalumab and up to 30 days after the last dose of durvalumab
* Patients receiving any chemotherapy, immunotherapy, biologic, radiotherapy or hormonal therapy for cancer treatment concurrently or within 3 weeks of study treatment. Concurrent use of hormonal therapy for non-cancer related conditions (e.g., hormone replacement therapy) is acceptable
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Participation in another clinical study with an investigational product administered in the last 3 months
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) or supportive care, while on the clinical study or during the follow-up period of this interventional study
* Patients with a known hypersensitivity to olaparib or durvalumab or any of the excipients of the product
* Involvement in the planning and/or conduct of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2025-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Durvalumab, Olaparib) - CDK12 and MMRd; Treatment (Durvalumab, Olaparib) - HRD: All patients receive durvalumab IV over 1 hour on day 1 of each cycle. Patients with CDK12 mutation and MMRd/MSI-high also receive olaparib PO BID on days 1- 28 of cycles 3-6. Patients with homologous recombination mutation also receive olaparib PO BID on days 1-28 of cycles 1-6. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Olaparib: Given PO
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Treatment (Durvalumab, Olaparib) - CDK12 and MMRd | Treatment (Durvalumab, Olaparib) - HRD
Started | 1 | 5
Completed | 1 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Durvalumab, Olaparib): All patients receive durvalumab IV over 1 hour on day 1 of each cycle. Patients with CDK12 mutation and MMRd/MSI-high also receive olaparib PO BID on days 1- 28 of cycles 3-6. Patients with homologous recombination mutation also receive olaparib PO BID on days 1-28 of cycles 1-6. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Olaparib: Given PO
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Note: All patients enrolled received combo therapy, so demographic data are provided in aggregate. Also, given the small number of enrolled subjects reporting demographics for the entire group is preferred.
Arm/Group | Treatment (Durvalumab, Olaparib)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Undetectable Prostate Specific Antigen (PSA)
Description: Will assess if patients achieve undetectable PSA for post-prostatectomy patients (including those that also received salvage radiation) or PSA < 0.5 ng/ml for post-definitive radiation patients.
Time Frame: At 12 months after initiation of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Durvalumab, Olaparib) - CDK12 and MMRd | Treatment (Durvalumab, Olaparib) - HRD
Number analyzed (Participants) | 1 | 5
Participants | 0 | 1

2. Secondary Outcome: PSA50 Response
Description: A descriptive summary (including the percentage and 90% confidence interval [CI]) of PSA50 response rate (proportion of patients with a decline in PSA > 50% from baseline) will be provided at 3- and 6-month timepoints. The response rate will be reported with exact binomial two-sided 90% CI.
Time Frame: At 3 and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Durvalumab, Olaparib) - CDK12 and MMRd | Treatment (Durvalumab, Olaparib) - HRD
Number analyzed (Participants) | 1 | 5
Participants | 0 | 3

3. Secondary Outcome: Change in Quality of Life: RANDSF-36
Description: RAND 36-Item Short Form (RANDSF-36) assesses physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, general health perceptions, and perceived change in health with a total score range of 0-100. The total score from all of the questions answered is divided by the total number of the questions answered yielding a global score from 0-100, with a higher score reflecting a better QoL. Mean difference in total average score is reported. Since the same treatment is used for all groups, we are reporting the data for RANDSF-36 in aggregate. Because this study terminated prematurely, the small number of enrolled subjects also preclude our ability to break this data at by subgroups.
Time Frame: At the time of enrollment and then every three months, with the last assessment at 12 months.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Treatment (Durvalumab, Olaparib) - HRD
Number analyzed (Participants) | 2
Scores on a scale | 4.64 [-1.14 to 10.42]

4. Secondary Outcome: Change in Quality of Life: IIEF
Description: International Index of Erectile Function (IIEF-5) is a diagnostic tool for erectile dysfunction, with a total score range of 5-25, with the lowest score indicating a higher degree of dysfunction. The mean difference in total score is reported. Since the same treatment is used for all groups, we are reporting the data for RANDSF-36 in aggregate. Because this study terminated prematurely, the small number of enrolled subjects also preclude our ability to break this data at by subgroups.
Time Frame: At the time of enrollment and then every three months, with the final measurement after 12 months.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Treatment (Durvalumab, Olaparib) - HRD
Number analyzed (Participants) | 2
Scores on a scale | -9 [-15 to -3]

ADVERSE EVENTS:
Time Frame: 90 days after the last dose of durvalumab or 30 days from last dose of olaparib, whatever comes later, up to 9 months. Note: Data is reported in aggregate since all patient received the same combination therapy. In addition, the small sample size due to early termination precludes breaking out the AEs by subgroup.
Arm/Group | Treatment (Durvalumab, Olaparib)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Durvalumab, Olaparib) (N=6)
Rash Pustular (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Durvalumab, Olaparib) (N=6)
Hot Flashes (Vascular disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT04336943/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT04336943/ICF_000.pdf